CLINICAL TRIAL: NCT04576637
Title: Neurophysiological Monitoring During Videolaryngoscopy and Tracheal Intubation in Patient With Unstable Cervical Spine: A Prospective, Interventional, Cohort Study
Brief Title: Neurophysiological Monitoring and Videolaryngoscopy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Leonid Eidelman, Professor Leonid Eidelman, Rabin Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 0534-20-RMC
Record Dates: First submitted 2020-09-22; First posted 2020-10-06 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-05

CONDITIONS: Postsynaptic Potential Summation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Neurophysiological monitoring during induction (Experimental)
  Interventions: Procedure: Neurophysiological monitoring during intubation

INTERVENTIONS:
Procedure: Neurophysiological monitoring during intubation — In the operating room patients will be connected to the anesthesia monitor and an IV line as standard clinical practice. Participants will receive oxygen and an IV infusion of 1-3 ng/ml remifentanil via TCI infusion pump to achieve mild sedation. Patients will then be connected to the neurophysiological electrodes to monitor for EEG, EMG, SSEP and MEP signals. After preparing the videolaryngoscope, anesthesia induction will be achieved with the use of IV ketamine 2mg/kg. Then the anesthesiologist will perform a clinical and ECG reading assessment to ensure that the patient is anesthetized and will be able to titrate more ketamine as needed to achieve hypnosis. A biteblock will be located to prevent teeth damage. A neurophysiological baseline recordings will then be performed by a neurophysiologist. The videolaryngoscope will then be inserted, during which a second neurophysiological testing will be performed to ensure the patients safety. Then mechanical ventilation will be initiated.

SUMMARY:
Myopathic patients undergoing cervical spine surgery are at risk for postoperative neurological deficits and sequelae.

Awake fiberoptic intubation is considered the technique of choice for tracheal intubation in patient with cervical spine instability. However, awake fiberoptic intubation frequently causes significant patient discomfort, requires patient cooperation, anesthesiologist expertise and the availability of costly equipment .

Videolaryngoscopy guided intubation is considered to be an effective alternative to awake fiberoptic intubation for cervical spine surgeries.

Intraoperative neurophysiological monitoring (IONM) is a method that provides real time evaluation of the functional integrity of neural structures. The goal of IONM is to make surgery safer by detecting incipient neurological insults at a time when it can be avoided or minimized and by aiding in the identification of neural structure Rayia, et al. have described a case of monitoring intubation and neck extension for the indication of thyroidectomy in a Down syndrome boy with atlantoaxial instability under anesthesia with propofol and remifentanil without neuromuscular blockade. The authors conclude that this approach can be used to protect against spinal cord compression.

While research has thoroughly evaluated the effect of laryngoscopy and intubation on cervical spine movement, to date, little is known about the impact of intubation process on neurophysiological responses, and on the feasibility of utilizing IONM for establishing a safe airway intubation.

This prospective, interventional, cohort study is the first, to our knowledge, to examine the feasibility and added benefits of IONM throughout anesthetic intubation in patients undergoing cervical spine surgeries with the use of videolarynscope guided intubation.

ELIGIBILITY:
Inclusion Criteria:

All patients above 18y old, presenting for cervical spine surgeries , suffering from cervical spine instability, whom are able to comply with the study requirements and gave a written informed consent will be eligible for study enrollment.

Exclusion Criteria:

* Patients presenting with heart disease will not be eligible to participate.
* Patients with anticipated difficult airway.
* Patients with a language barrier.
* Patients with known allergy to any of the drugs used.
* Pregnant women
* Patients with a history of seizures or CVA.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-10-21 (Actual); Primary Completion 2022-12-21 (Estimated); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Differences is somatosensory evoked potentials and motor evoked potentials signals during intubation | During surgery

CONTACTS AND LOCATIONS:
Overall Officials: Leonid O Eidelman, Principal Investigator — Rabin Medical Center
Locations (1):
- Rabin Medical Center/Beilinson Campus, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Epstein NE. The need to add motor evoked potential monitoring to somatosensory and electromyographic monitoring in cervical spine surgery. Surg Neurol Int. 2013 Oct 29;4(Suppl 5):S383-91. doi: 10.4103/2152-7806.120782. eCollection 2013. PMID 24340237
- [Background] Dutta K, Sriganesh K, Chakrabarti D, Pruthi N, Reddy M. Cervical Spine Movement During Awake Orotracheal Intubation With Fiberoptic Scope and McGrath Videolaryngoscope in Patients Undergoing Surgery for Cervical Spine Instability: A Randomized Control Trial. J Neurosurg Anesthesiol. 2020 Jul;32(3):249-255. doi: 10.1097/ANA.0000000000000595. PMID 30925539
- [Background] Stecker MM. A review of intraoperative monitoring for spinal surgery. Surg Neurol Int. 2012;3(Suppl 3):S174-87. doi: 10.4103/2152-7806.98579. Epub 2012 Jul 17. PMID 22905324
- [Background] Nunes RR, Bersot CDA, Garritano JG. Intraoperative neurophysiological monitoring in neuroanesthesia. Curr Opin Anaesthesiol. 2018 Oct;31(5):532-538. doi: 10.1097/ACO.0000000000000645. PMID 30020157
- [Background] Al Bahri RS, MacDonald DB, Mahmoud AH. Motor and somatosensory evoked potential spinal cord monitoring during intubation and neck extension for thyroidectomy in a Down syndrome boy with atlantoaxial instability. J Clin Monit Comput. 2017 Feb;31(1):231-233. doi: 10.1007/s10877-016-9832-x. Epub 2016 Jan 28. PMID 26820847